CLINICAL TRIAL: NCT04650178
Title: COVID-19: Well-Being in Cancer Patients With Neuropathy Who Participated in Prior Clinical Trials
Brief Title: Well-being in Cancer Patients With Neuropathy During COVID-19 Who Participated in Prior Clinical Trials
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0508; NCI-2020-06014 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0508 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-19; First posted 2020-12-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Neuropathy
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, quality of life): Patients complete an online questionnaire over 15 minutes about their experiences regarding the COVID-19 pandemic including testing, risks of exposure, whether people they know have acquired COVID-19, as well as questions on how the pandemic has impacted their quality of life.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study investigates the experiences of cancer patients with neuropathy during the COVID-19 pandemic to learn how the COVID-19 pandemic affects their quality of life and clinical outcomes. This study will also explore whether there are differences between patients who received neurofeedback (NFB, a type of therapy that is thought to help normalize brain activity) and those who did not. Learning about quality of life in cancer patients with neuropathy during the COVID-19 pandemic may help guide development of programs and policies to improve chronic pain patient care and outcomes during a major global healthcare crisis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess experiences during the coronavirus disease 2019 (COVID-19) pandemic of the health-related quality of life (HRQOL) (e.g. physical, emotional, social well-being), and other COVID-19-specific domains (e.g. anxiety, social interactions, finances), and the associations between COVID-19 experiences and COVID-19-specific distress, HRQOL and clinical outcomes of patients who participated in one of three clinical trials.

II. Examine differences in outcomes between neuropathic pain patients who participated in one of two trials of NFB and received NFB, and neuropathic pain patients who participated in a non-treatment-related neuropathy study (i.e., who did not receive NFB).

III. Evaluate the extent to which coping and resilience factors moderate the effects of COVID-19 experiences on COVID-19-specific distress, HRQOL and clinical outcomes.

OUTLINE:

Patients complete an online questionnaire over 15 minutes about their experiences regarding the COVID-19 pandemic including testing, risks of exposure, whether people they know have acquired COVID-19, as well as questions on how the pandemic has impacted their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in one of the following protocols: 2015-0399, 2012-0642, or 2010-0675
* Has an active email address or can be contacted by MyChart or personal email

Exclusion Criteria:

* No evidence of consent from prior clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients with neuropathy who have participated in one of the following clinical trials: 2015-0399, 2012-0642, or 2010-0675.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life and coronavirus disease 2019 (COVID-19)-specific domains of interest | through study completion, an average of 6 months
  We will use the COVID-19 Specific questionnaire. This scale will ask 15 questions that are organized into three sections: (a) Questions specific to the COVID-19 pandemic such as testing, serostatus, risk factors, loss of family or friends, isolation; (b) Thoughts, experiences and emotions regarding the COVID-19 pandemic; and (c) Health-related quality of life. This assessment was developed by Lorenzo Cohen (MD Anderson), in collaboration with investigators from the University of Miami and UCLA and is a comprehensive assessment of COVID-19 experiences.
COVID-19 experiences and COVID-19 specific distress | through study completion, an average of 6 months
  Will evaluate bivariate associations between COVID-19 experiences and COVID-19-specific distress, HRQOL and clinical outcomes, using Pearson product-moment correlation coefficients, chi-squared tests, or analyses of variance (ANOVA) where appropriate.
Differences in outcomes between neuropathic pain patients | through study completion, an average of 6 months
  Will use linear regression (or generalized linear models, as applicable) to assess differences in the outcomes of interest between neuropathic pain patients who received neurofeedback (NFB) from either of the two NFB trials (principal investigator [PI]: Dr. Prinsloo) and the neuropathic pain patients who participated in Dr. Gibby-Reyes' trial (who, consequently, did not receive NFB).
Coping and resilience factors | through study completion, an average of 6 months
  Will preliminarily test the interaction effect between each of the coping and resilience factors and COVID-19 experiences on COVID-19-specific distress, HRQOL and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org